CLINICAL TRIAL: NCT04920916
Title: Safety and Efficacy of the Treatment of Hospitalized Patients With COVID 19 Infection With an Inhibitor of IL-4 and IL-13 Signaling: A Phase IIa Trial
Brief Title: Safety and Efficacy of Dupilumab for Treatment of Hospitalized COVID-19 Patients
Acronym: SafeDrop
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: The Paul Manning Foundation (Other); Virginia Catalyst (Other)
Responsible Party: Principal Investigator, William Petri, MD, PhD, Wade Hampton Frost Professor of Medicine and Vice Chair for Research of the Department of Medicine, and Professor of Medicine, Microbiology, Immunology and Cancer Biology, and Pathology, Medicine: Infectious Diseases and International Health, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSR210184; HSR220171 (Other: UVA IRB)
Record Dates: First submitted 2021-06-08; First posted 2021-06-10 (Actual); Results first posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: COVID-19
Keywords: Anti-Inflammatory Agents
MeSH Terms: conditions — COVID-19 | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dupilimab (Experimental): Dupilimab: 600 mg, given as two 300 mg subcutaneous injections on day 0/1. If participants are still hospitalized a second and third dose (300 mg) will be given on days 14 and 28.
  Interventions: Biological: Dupilumab
- Placebo (Placebo Comparator): Normal saline will be given as two one mL subcutaneous injections on day 0/1. If participants are still hospitalized a second and third dose (1 mL) will be given on days 14 and 28.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Dupilumab — Participants will receive a loading dose of dupilumab (600 mg, given as two 300 mg subcutaneous injections) on day 0/1. If participants are still hospitalized a second and third dose (300 mg) will be given on days 14 and 28.
  Other Names: Dupixent
  Arms: Dupilimab
Drug: Placebo — Normal Saline.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, superiority phase IIa trial to assess the safety and efficacy of dupilumab use in hospitalized patients with moderate to severe COVID-19 infection. Subsequently, we conducted a 1 year follow up study to investigate the occurrence of Post COVID conditions (PCC) in our study population through assessment of pulmonary function, symptoms, neurocognition and immune biomarkers to observe for any treatment group differences.

DETAILED DESCRIPTION:
A total of 40 eligible subject were enrolled and randomized in a 1:1 ratio to receive either dupilumab or placebo, stratifying on the disease severity measured by the required oxygen ≤ 15L or > 15L by nasal cannula. Both arms received standard of care management per current National Institutes of Health (NIH) COVID-19 treatment guideline in addition to their randomized treatments. Patients were then followed prospectively for up to 360 days after enrollment.

As an extension to the randomized double-blind placebo-controlled trial assessing dupilumab for treatment of those hospitalized with acute moderate to severe COVID-19, subjects were followed up at 1 year for evaluation of pulmonary function testing (PFT), pulmonary imaging, immune biomarkers, neurocognition and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older at the time of enrollment.
* Patients hospitalized with a positive RT-PCR for SARS-CoV-2 within the last 14 days, with illness duration within the last 14 days, and evidence of moderate to severe COVID-19 infection as defined by NIH COVID-19 Severity Categorization (8):

  * Moderate illness: Individuals who show evidence of lower respiratory disease during clinical assessment or imaging and who have saturation of oxygen SpO2≥ 94% on room air at sea level.
  * Severe illness: Individuals who have SpO2 <94% on room air at sea level, a ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mm Hg, respiratory frequency >30 breaths/min, or lung infiltrates >50%.
* Patient and/or legally authorized representative is willing and able to provide written informed consent and comply with all protocol requirements.
* Patients with hematologic malignancies or solid tumors are eligible.
* Patients with autoimmune disorders are eligible.
* Patients with immunodeficiency and organ or stem cell transplant recipients are eligible.
* Patients with acute or chronic renal injury/failure are eligible.
* Patients with neutropenia/lymphopenia are eligible.
* Patients with elevated liver function tests are eligible.
* Women who are not taking contraception are eligible.
* Patients who are currently or have recently received steroids and/or remdesivir are eligible.
* Patient agrees to not participate in another clinical trial for the treatment of COVID-19 through end of study period.

Exclusion Criteria:

* Patients who do not require inpatient admission for COVID-19 infection.
* Patients who require invasive mechanical ventilation at time of enrollment.
* A pre-existing condition or use of a medication that, in the opinion of the site investigator, may place the individual at a substantially increased risk due to study participation.
* Pregnancy or breast feeding (lactating women who agree to discard breast milk from day 1 until two weeks after the last study product is given are not excluded).
* Allergy to Dupilumab or its excipients.
* Received any of the following in the two weeks prior to screening as treatment of COVID-19:
* small molecule tyrosine kinase inhibitors (e.g. imatinib, gefitinib, acalabrutinib, etc.);
* monoclonal antibodies targeting cytokines (e.g., TNF inhibitors, anti-interleukin-1 [IL-1], anti-IL-6 [or sarilumab], etc.);
* monoclonal antibodies targeting T-cells or B-cells as treatment for COVID-19;
* Any other immunomodulatory (other than steroids) medications within 5 half-lives or 30 days prior to randomization.
* Current acute parasitic helminth infection or history of chronic parasitic infection.
* History of ocular scleritis, uveitis, keratitis or recent (<6 months) eye injury (chemical or traumatic), infection or vascular occlusion.
* Have received any live vaccine (that is, live attenuated) within 4 weeks before screening, or intend to receive a live vaccine (or live attenuated) during the study. Note: Use of non-live (inactivated) vaccinations is allowed for all subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William A Petri Jr., MD, PhD, Principal Investigator — University of Virginia Division of Infectious Disease
Locations (1):
- UVA Health, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Sasson J, Donlan AN, Ma JZ, Haughey HM, Coleman R, Nayak U, Mathers AJ, Laverdure S, Dewar R, Jackson PEH, Heysell SK, Sturek JM, Petri WA Jr. Safety and Efficacy of Dupilumab for the Treatment of Hospitalized Patients With Moderate to Severe Coronavirus Disease 2019: A Phase 2a Trial. Open Forum Infect Dis. 2022 Jul 27;9(8):ofac343. doi: 10.1093/ofid/ofac343. eCollection 2022 Aug. PMID 35959207
- [Result] Hendrick J, Ma JZ, Haughey HM, Coleman R, Nayak U, Kadl A, Sturek JM, Jackson P, Young MK, Allen JE, Petri WA Jr. Pulmonary function and survival one year after dupilumab treatment of acute moderate to severe COVID-19: A follow up study from a Phase IIa trial. medRxiv [Preprint]. 2023 Sep 2:2023.09.01.23293947. doi: 10.1101/2023.09.01.23293947. PMID 37693596
- [Derived] Sasson J, Donlan AN, Ma JZ, Haughey HM, Coleman R, Nayak U, Mathers AJ, Laverdure S, Dewar R, Jackson PEH, Heysell SK, Sturek JM, Petri WA Jr. Safety and Efficacy of Dupilumab for the Treatment of Hospitalized Patients with Moderate to Severe COVID 19: A Phase IIa Trial. medRxiv [Preprint]. 2022 May 19:2022.03.30.22273194. doi: 10.1101/2022.03.30.22273194. PMID 35411349

RESULTS

PARTICIPANT FLOW:
Groups:
- Dupilimab: Active Dupilimab: 600 mg, given as two 300 mg subcutaneous injections on day 0/1. If participants are still hospitalized a second and third dose (300 mg) will be given on days 14 and 28.
  Dupilumab: Participants will receive a loading dose of dupilumab (600 mg, given as two 300 mg subcutaneous injections) on day 0/1. If participants are still hospitalized a second and third dose (300 mg) will be given on days 14 and 28.
- Placebo: Dupilimab Placebo: placebo (normal saline) will be given as two one mL subcutaneous injections on day 0/1. If participants are still hospitalized a second and third dose (1 mL) will be given on days 14 and 28.
  Placebo: Participants will receive a loading dose of normal saline (2 ml, given as two one ml subcutaneous injections) on day 0/1. If participants are still hospitalized a second and third dose (1 ml) will be given on days 14 and 28.
Period: Phase IIa 60 Day Study
Arm/Group | Dupilimab | Placebo
Started | 19 | 21
Completed | 17 | 16
Not Completed | 2 | 5
Not completed — Death | 2 | 5
Period: 1 Year Follow up (Phone Call)
Arm/Group | Dupilimab | Placebo
Started | 17 | 16
Completed | 16 | 13
Not Completed | 1 | 3
Not completed — Death | 1 | 3
Period: 1 Year Follow up Visits
Arm/Group | Dupilimab | Placebo
Started | 16 | 13
Completed | 10 | 6
Not Completed | 6 | 7
Not completed — Lost to Follow-up | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Dupilimab: Participants will receive a loading dose of dupilumab (600 mg, given as two 300 mg subcutaneous injections) on day 0/1. If participants are still hospitalized a second and third dose (300 mg) will be given on days 14 and 28.
- Placebo: Participants will receive a loading dose of normal saline (2 ml, given as two one ml subcutaneous injections) on day 0/1. If participants are still hospitalized a second and third dose (1 ml) will be given on days 14 and 28.
- Total: Total of all reporting groups
Arm/Group | Dupilimab | Placebo | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [33 to 85] | 63 [40 to 86] | 61.5 [38.5 to 84.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 7 | 16 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 16 | 18 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 19 | 21 | 40
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 33.6 [18.7 to 48.5] | 32.3 [22.2 to 42.4] | 33 [22.7 to 43.3]

OUTCOME MEASURES:

1. Primary Outcome: Day 28 Ventilator Free Survival
Description: Proportion of patients alive and free of invasive mechanical ventilation
Time Frame: at 28 Days ± 2d
Measure: Number; unit: proportion of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 19 | 21
proportion of participants | 0.79 | 0.86

2. Primary Outcome: Follow up Study 1 Year Outcome: Pulmonary Function Testing- Oxygen Diffusion and 6 Minute Walk Testing
Description: Proportion of patients with abnormal diffusing capacity for carbon monoxide (DLCO) and/or 6 minute walk testing 1 year after acute COVID-19 infection.
Time Frame: 365 ± 90 days
Measure: Number; unit: proportion of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 10 | 6
proportion of participants | 0.30 | 1.0

3. Secondary Outcome: Proportion of Patients With Eosinophilia
Description: defined as an absolute eosinophil count > 0.6 k/µl at ≥ 1 measurement throughout the study period
Time Frame: Day 0 through Day 60
Measure: Number; unit: proportion of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 19 | 21
proportion of participants | 0.26 | 0.048

4. Secondary Outcome: Cumulative Incidence of Grade 3 and 4 Clinical Adverse Events, Serious Adverse Events (SAEs) or Death
Description: defined as number of new events divided by the total number of individuals in the population at risk for the time interval
Time Frame: Day 0 through Day 60
Measure: Number; unit: percent of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 19 | 21
percent of participants | 58 | 29

5. Secondary Outcome: SARS-CoV-2 Variants
Description: Prevalence of delta variant in study population.
Time Frame: Day 0
Population: Five and four samples from the placebo and dupilumab groups, respectively, were unable to undergo sequencing.
Measure: Number; unit: percentage of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 15 | 16
percentage of participants | 100 | 94

6. Secondary Outcome: Change in Plasma Total Immunoglobulin E (IgE) Levels
Description: Change in levels (difference between day 14- day 0 levels).
Time Frame: Day 0 and Day 14
Population: Two subjects in the both the dupilumab and placebo groups were unable to undergo day 14 IgE assessment.
Measure: Median (Inter-Quartile Range); unit: U/mL
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 17 | 19
U/mL | 17.5 [6.1 to 53.8] | 16.3 [2.6 to 81.0]

7. Secondary Outcome: Change in C-reactive Protein (CRP)
Description: Change in levels (difference between day 14- day 0 levels)
Time Frame: Day 0 through Day 14
Population: One and two patients in the placebo and dupilumab groups, respectively, were unable to undergo day 14 CRP assessment.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 17 | 20
mg/dL | 5.5 [2.3 to 14.3] | 8.9 [4.95 to 10.1]

8. Secondary Outcome: Change in Ferritin
Description: Change in levels (difference between day 14- day 0 levels).
Time Frame: Day 0 through Day 14
Population: One and two patients in the placebo and dupilumab groups, respectively, were unable to undergo day 14 ferritin level assessment.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 17 | 20
ng/mL | 384 [131 to 595] | 545 [10.5 to 1115.5]

9. Secondary Outcome: Duration of Hospitalization
Description: Measured in days
Time Frame: Day 0 through Day 30
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 19 | 21
days | 6 [4 to 22] | 6 [5 to 18]

10. Secondary Outcome: Day 60 All Cause Mortality
Description: All cause mortality by day 60
Time Frame: Day 60
Measure: Number; unit: percentage of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 19 | 21
percentage of participants | 11 | 24

11. Secondary Outcome: Day 28 All-cause Mortality Rate
Description: Mortality rate
Time Frame: at Day 28
Measure: Number; unit: percentage of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 19 | 21
percentage of participants | 5 | 14

12. Secondary Outcome: Day 60 Ventilator Free Survival
Description: Proportion of patients alive and free of invasive mechanical ventilation
Time Frame: Day 60
Measure: Number; unit: proportion of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 19 | 21
proportion of participants | 0.90 | 0.76

13. Secondary Outcome: Percentage of Patients Needing Extracorporeal Membrane Oxygenation (ECMO)
Description: Percentage
Time Frame: Day 0 through Day 60
Measure: Number; unit: percentage of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 19 | 21
percentage of participants | 0 | 0

14. Secondary Outcome: Percentage of Patients Needing Renal Replacement Therapy
Description: Percentage
Time Frame: Day 0 through Day 60
Measure: Number; unit: percentage of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 19 | 21
percentage of participants | 11 | 10

15. Secondary Outcome: Percentage of Patients Needing Vasopressors
Description: Percentage
Time Frame: Day 0 through Day 60
Measure: Number; unit: percentage of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 19 | 21
percentage of participants | 21 | 19

16. Secondary Outcome: Follow Up Study 1 Year Outcome: All-cause Mortality at 1 Year
Description: Percent of subjects who died by 1 year.
Time Frame: 365 days
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Dupilimab Placebo: placebo (normal saline) will be given as two one mL subcutaneous injections on day 0/1. If participants are still hospitalized a second and third dose (1 mL) will be given on days 14 and 28.
  Placebo: Normal Saline.
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 19 | 21
percentage of participants | 16 | 38

17. Secondary Outcome: Follow-up Study 1 Year Outcome: Differences in High Resolution Computed Tomography (HRCT) Chest Scan Appearance Post Recovery
Description: Compare Enrollment HRCT to 1 year HRCT. Percent of abnormal on CT. Reported as percent of subjects with any abnormality on CT.
Time Frame: 365 ± 90 days
Measure: Number; unit: Percentage of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 10 | 6
Percentage of participants | 80 | 67

18. Secondary Outcome: Follow-up Study 1 Year Outcome: Conduct a 6 Minute Walk Testing
Description: Proportion of patients with greater than 3% oxygen desaturation during 6 minute walk testing
Time Frame: 365 ± 90 days
Measure: Number; unit: Proportion of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 10 | 6
Proportion of participants | 0.10 | 0.50

19. Secondary Outcome: Follow up Study 1 Year Outcome: Pulmonary Function Testing- Abnormal Spirometry
Description: Percentage of subjects with a percent of predicted (compared to Global Lung Function Initiative (GLI) predicted values based on age, sex, height and ethnicity) below normal for forced expiratory volume (FEV1) or forced vital capacity (FVC), which are measures used to determine the volume of air that can be exhaled in one breath.
Time Frame: 365 ± 90 days
Measure: Number; unit: percentage of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 10 | 6
percentage of participants | 30 | 67

20. Secondary Outcome: Follow-up Study 1 Year Outcome: Assess Neurocognitive Function Using the MOCA
Description: Determine the proportion of patients with reduce neurocognitive function. Neurocognitive testing included completion of Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety, PROMIS Depression, the Montreal Cognitive Assessment (MOCA), the Insomnia Severity Index (ISI), the Katz Index of Independence In Activities of Daily Living (Katz-ADL), EuroQOL (EQ)-5D-5L and Neuro- Quality of Life (QoL) questionnaires. Reduced neurocognitive function was determined if scoring from at least one of these tests was deemed a variation from population norm per scoring instructions.
Time Frame: 365 ± 90 days
Measure: Number; unit: proportion of participants
Arm/Group | Dupilimab | Placebo
Number analyzed (Participants) | 10 | 6
proportion of participants | 0.90 | 0.83

ADVERSE EVENTS:
Time Frame: Adverse events were collected on study day 0, 2, 5, 7, 14, 28 and 60 in initial Phase IIa study. Day 7, 28 and 60 were considered optional, although recommended, if patient discharged within the time frame. No SAEs/AEs were collected past day 60. Therefore, while all cause mortality was assessed up to 1 year, other AEs/SAEs were assessed up to day 60.
Description: All cause mortality was assessed up to 1 year. Other AEs/SAEs were assessed only up until day 60.
Arm/Group | Dupilimab | Placebo
All-Cause Mortality (participants affected / at risk) | 3/19 | 8/21
Serious Adverse Events (participants affected / at risk) | 11/19 | 6/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dupilimab (N=19) | Placebo (N=21)
Injection Site Reactions (Injury, poisoning and procedural complications) | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 2
Bacterial pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Herpes viral infection (Infections and infestations) | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 5 | 1
Hypereosinophilic syndrome (Immune system disorders) | 0 | 0
Other infections (Infections and infestations) | 4 | 2 — Other infections included Clostridioides difficile infection (1), bacteremia (2), urinary tract infections (2) and oral candidiasis (1).

LIMITATIONS AND CAVEATS:
This was a small study, designed as an early phase trial. Limitations included lack of achievement of the primary endpoint and the wide confidence intervals in the survival benefit of dupilumab at day 60. Additional limitations included unequal gender distribution between groups (also due to small sample size), patients were almost exclusively infected by the Delta variant of SARS CoV-2 and a higher-than-expected overall mortality rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol: Phase IIa Study (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT04920916/Prot_003.pdf
  • Study Protocol: 1 year follow up of Phase IIa study (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT04920916/Prot_004.pdf
  • Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT04920916/SAP_002.pdf